CLINICAL TRIAL: NCT04149223
Title: Cirrhosis Care Alberta (CCAB): A Pragmatic Type II Hybrid Effectiveness Implementation Trial Evaluating the Effectiveness of a Standardized Order Set
Brief Title: Cirrhosis Care Alberta (CCAB): A Pragmatic Type II Hybrid Effectiveness Implementation Trial
Acronym: CCAB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Alberta Innovates Health Solutions (Other); Alberta Health services (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro000089501
Record Dates: First submitted 2019-08-12; First posted 2019-11-04 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Cirrhosis, Liver
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Intervention Model Description: The experimental design is a stepped roll-out hybrid II effectiveness-implementation trial (Curran et al. 2012), which tests clinical intervention impact and rigorously evaluates implementation strategy in real time. Over three years, the investigators will implement the CCAB intervention across 8 Alberta hospital sites within Alberta Health Services (AHS). The overarching objective of this study is to demonstrate both effectiveness and implementation feasibility for routine patient care within AHS.
  Given the pragmatic approach to this study, the commencement and scale-up of the study will coincide with the phases of the planned roll-out of Connect Care (the new Alberta Electronic Medical Record (EMR) platform) across the province. The project allows for an incredibly interesting and unique opportunity to implement and evaluate a comprehensive provincial chronic disease intervention in a real-world context, both in current state and with EMR facilitation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Current practice at baseline, routine cirrhosis care.
- Intervention (Experimental): Use of a standardized cirrhosis order set.
  Interventions: Other: Evidence-based standardized Cirrhosis order set
- Intervention + EMR (Active Comparator): Use of a standardized cirrhosis order set embedded within an electronic medical record.
  Interventions: Other: Evidence-based standardized Cirrhosis order set

INTERVENTIONS:
Other: Evidence-based standardized Cirrhosis order set — Standardized order sets for guidance in ascites, varices, hepatic encephalopathy, infections, and medication reconciliation (optimizing HE medication, medication prophylaxis, withdrawal of non-indicated proton pump inhibitors).
  Arms: Intervention; Intervention + EMR

SUMMARY:
Liver cirrhosis is the leading cause of morbidity and premature mortality in patients with digestive disease. There are many gaps in care which contribute to a high rate of hospital readmissions (44 percent at 90 days) and inadequate quality of care. Currently, there is a lack of structured processes to initiate best practice support for medical and broader health needs of high risk patients.

The cirrhosis care Alberta program (CCAB) is a 3 year multi-component quality improvement initiative which will aim to improve quality of care, reduce acute care utilization and be satisfactory to both patients and providers. Best practice support will be provided in the areas of: Evidence based management of cirrhosis, alcohol use support, frailty, advance care planning, home-hospital-home transitions including standardized outpatient monitoring and structured urgent access for rapid, on-demand outpatient assessment.

DETAILED DESCRIPTION:
Cirrhosis Care Alberta (CCAB) is a 3 year multi-component system-wide quality improvement trial which aims to improve quality of care, reduce acute care utilization and meet the needs of both patients and providers throughout Alberta. Instead of addressing just a single contributor to acute care utilization, this ambitious intervention will be the first in the world to bring together care providers across the province to tackle the complex multilevel problem with a multilevel solution. The intervention includes implementation of our standardized integrated strategy for delivering evidence-based best practices under real-world conditions to address the key determinants of hospital readmission and length of stay (LOS) in patients admitted with cirrhosis.

The CCAB project intervention includes:

1. Comprehensive Care Bundle (development underway):

   1. Admission and Discharge/Transition order set focused on the screening and management of:

      * Cirrhosis complications
      * Frailty and malnutrition
      * Alcohol use disorder and
      * Transition to community
   2. Patient and caregiver education

      • A major theme that came up in focus group work with patients and in the literature is the lack of useful information that is available to them. This is a top priority for patients. Education will include guidelines and tools for patients to improve self-management as well as support for caregivers.
   3. Provider education

      * Nursing education focused on providing teaching to patients with cirrhosis and initiating alcohol screening and performing a brief intervention to promote abstinence is done in the minority of patients at discharge.
      * Physician education focused on cirrhosis complications and broader health needs such as prescribing pharmacological therapies for alcohol use disorder (currently done in <5% of patients even though the number needed to treat is 12 (i.e. need to do it in 12 patients to result in a benefit)).
2. Community Care Pathways

   1. Hepatic Encephalopathy (HE) Pathway: HE is the most common reason for admission to hospital and is a significant burden on patients and families. In collaboration with Health Link, this project aims to develop a call pathway so that patients and families can receive best practice support by nurses in the community and avoid needing to access emergency departments when HE can safely be managed in the community. The patient education surrounding HE is being developed as part of the Care Bundle, but developing a care pathway will ensure the education is translated and reinforced.
   2. Ascites Pathway: Ascites (abdominal fluid build-up) is the most common cirrhosis related complication and is extremely uncomfortable for patients. When diuretics are not tolerated or ineffective, this population typically requires frequent draining of the ascites fluid (paracentesis) to treat symptoms such as shortness of breath, pain and inability to eat. Paracentesis is usually performed in hospital based day procedure areas, but when patients can not access a scheduled paracentesis in a timely manner, they are left with no option other than going to emergency rooms. Through process mapping and identifying current barriers and facilitators with each site, the project team aims to develop effective pathways for linking patients in with timely paracentesis.

ELIGIBILITY:
Inclusion Criteria:

* Adults (great than 18 years of age) with a clinical diagnosis of cirrhosis (confirmed by compatible radiology, histology or fibroscan)
* Admitted to a study hospital site

Exclusion Criteria

o Adult patients who do not have cirrhosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3975 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Cumulative hospital length of stay (LOS) per patient year | Baseline, 1 year, 2 year
  LOS

SECONDARY OUTCOMES:
Hospital Readmission Rate | Baseline,through study completion, an average of 1 year
  Readmission rate
Mean Length of Stay (LOS) (Ward, ICU, Total) | Baseline,through study completion, an average of 1 year
  LOS
Readmission rate at 90 days | From commencement of the study (baseline), assessed quarterly until study completion.
  Readmission rate
Emergency Department (ED) Visit Rate | Baseline,through study completion, an average of 1 year
  ED visit rate
Outpatient Visit rate | Baseline,through study completion, an average of 1 year
  by provider type, location
Survival | Baseline,through study completion, an average of 1 year
  Patient with cirrhosis survival
Disease severity | Baseline,through study completion, an average of 1 year
  laboratory values, model for end-stage liver disease (MELD) score
Implementation fidelity | From commencement of the study (baseline), assessed quarterly until study completion.
  Adherence to cirrhosis order set

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carbonneau M, Eboreime EA, Hyde A, Campbell-Scherer D, Faris P, Gramlich L, Tsuyuki RT, Congly SE, Shaheen AA, Sadler M, Zeman M, Spiers J, Abraldes JG, Sugars B, Sia W, Green L, Abdellatif D, Schaefer JP, Selvarajah V, Marr K, Ryan D, Westra Y, Bakshi N, Varghese JC, Tandon P. The cirrhosis care Alberta (CCAB) protocol: implementing an evidence-based best practice order set for the management of liver cirrhosis - a hybrid type I effectiveness-implementation trial. BMC Health Serv Res. 2020 Jun 18;20(1):558. doi: 10.1186/s12913-020-05427-8. PMID 32552833